CLINICAL TRIAL: NCT05525611
Title: Cabergoline as a Preventive Treatment for Chronic Migraine: an Investigator-Initiated, Randomized Clinical Trial
Brief Title: Cabergoline as a Preventive Treatment for Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Migraine_2022
Record Dates: First submitted 2022-06-01; First posted 2022-09-01 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2022-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Cabergoline

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled parallel study with a 12 weeks duration.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabergoline (Experimental)
  Interventions: Drug: Cabergoline 0.5 MG
- Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cabergoline 0.5 MG — Cabergoline 0.5 mg once a week in 12 weeks
  Arms: Cabergoline
Other: Placebo — Placebo once a week in 12 weeks
  Arms: Control

SUMMARY:
Headache disorders constitute a major global disease burden, and migraine - with a one-year prevalence of 15 % - is the sixth most disabling condition. Though a common disease, the pathogenesis is still unclear. Thus, the treatments have different mechanisms of action and preventive treatments are only effective in approximately 50% of chronic migraine patients. Recent evidence from mice models and a study of prolactine-associated headaches have indicated that dopamine agonists such as cabergoline might be used as a treatment of migraine.

The aim of this study is to test the hypothesis that the dopamine agonist cabergoline can be used as a treatment of chronic migraine. A randomized controlled trial of 24 patients with chronic migraine will be conducted, comparing cabergoline to placebo as an add-on medication to the patients' migraine treatment over a 12 weeks period. The primary outcome is change in migraine frequency, but also headache-related hospital contacts, and quality of life as well as prolactin levels and biomarkers of the pituitary-gonadal-axis. The results of the study will help understand the pathogenesis of migraine and might also introduce a more effective and affordable preventive migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Migraine and more than 6 days with headache every months

Exclusion Criteria:

* Cardiac valve disease
* Hypertension
* Psychiatric disease
* Treated with dopamine receptor agonists, dopamin receptor antagonists, macrolides and itraconazole
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
A change in days with headache in patients with chronic migraine | 12 weeks
  Based on a headache diary

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Laboratory, Department of Clinical Medicine, Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus N, Central Jutland, Denmark

REFERENCES:
- [Derived] Hjelholt AJ, Bach FW, Kasch H, Stovring H, Jensen TS, Jorgensen JOL. Cabergoline as a preventive migraine treatment: A randomized clinical pilot trial. PLoS One. 2025 Apr 1;20(4):e0320937. doi: 10.1371/journal.pone.0320937. eCollection 2025. PMID 40168298